CLINICAL TRIAL: NCT06459297
Title: Post-marketing Surveillance to Evaluate the Safety and Effectiveness of Upadacitinib (RINVOQ) in Korean Adult Patients With Ulcerative Colitis or Crohn's Disease
Brief Title: Study of Oral Upadacitinib to Assess Change in Disease Activity and Adverse Events in Adult Participants With Ulcerative Colitis or Crohn's Disease
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-081
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Inflammatory Bowel Diseases; Upadacitinib; RINVOQ; Ulcerative colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Upadacitinib: Participants will receive upadacitinib as prescribed by their physician according to local label.

SUMMARY:
Ulcerative colitis (UC) is an idiopathic, chronic, inflammatory disease affecting the colon. Crohn's disease (CD) is an incurable chronic inflammatory disorder of the gastrointestinal tract. This study will assess how safe and effective upadacitinib is in treating adult participants with moderate to severe ulcerative colitis and Crohn's disease. Adverse events and change in disease activity will be assessed.

Upadacitinib is an approved drug for treating Atopic dermatitis (AD), psoriatic arthritis (PsA), ankylosing spondylitis (AS), non-radiographic axial spondyloarthritis (nr-axSpA), ulcerative colitis (UC), and Crohn's disease (CD). Approximately 600 adult participants who are prescribed Upadacitinib by their physician in accordance with local label will be enrolled in Korea.

Upadacitinib will be administered in accordance with the terms of the local marketing authorization, and treatment of participants will be determined solely by the investigator. Participants in the study will be followed for up to 52 weeks.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosis with ulcerative colitis or Crohn's Disease suitable for the treatment with Upadacitinib.
* Participants prescribed upadacitinib in accordance with the approved local label.

Exclusion Criteria:

* Participants with any contraindication to Upadacitinib.
* Participants currently participating in another clinical research not including observational study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with ulcerative colitis or Crohn's Disease
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who reported Serious Adverse Event | Up to 52 weeks
  An Adverse Event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Percentage of participants who reported Serious Adverse Drug Reaction | Up to 52 weeks
  An Adverse Event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment. Among AEs, an event whose causal relationship with the product cannot be ruled out is considered an adverse drug reaction.
Percentage of participants who reported unexpected (not reflected in the latest approved label) Adverse Events/Adverse Drug Reaction | Up to 52 weeks
  An Adverse Event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment. Among AEs, an event whose causal relationship with the product cannot be ruled out is considered an adverse drug reaction.
Percentage of participants who reported known (labeled) Adverse Drug Reaction | Up to 52 weeks
  An Adverse Event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment. Among AEs, an event whose causal relationship with the product cannot be ruled out is considered an adverse drug reaction.
Percentage of participants who reported non-serious Adverse Event/Adverse Drug Reaction | Up to 52 weeks
  An Adverse Event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment. Among AEs, an event whose causal relationship with the product cannot be ruled out is considered an adverse drug reaction.
Percentage of participants who reported the events related to important identified risks/important potential risks/missing information | Up to 52 weeks
  An Adverse Event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment. Among AEs, an event whose causal relationship with the product cannot be ruled out is considered an adverse drug reaction.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (14):
- South Korea (14):
  - SoonChunHyang University Hospital Cheonan /ID# 270015, Cheonan-si, Chungcheongnam-do
  - The Catholic University of Korea, Daejeon St. Mary's Hospital /ID# 267843, Daejeon, Daejeon Gwang Yeogsi
  - Inje University - Ilsan Paik Hospital /ID# 269995, Goyang-si, Gyeonggido
  - Keimyung University Dongsan Hospital /ID# 269775, Daegu, Gyeongsangbuk-do
  - Chosun University Hospital /ID# 269990, Gwangju, Jeonranamdo
  - Kyung Hee University Hospital /ID# 270003, Dongdaemun-gu, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 268865, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital /ID# 270020, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 270014, Seoul, Seoul Teugbyeolsi
  - Hallym University Kangnam Sacred Heart Hospital /ID# 270013, Seoul, Seoul Teugbyeolsi
  - Ewha Womans University Medical Centre /ID# 269776, Seoul, Seoul Teugbyeolsi
  - Ulsan University Hospital /ID# 270006, Ulsan, Ulsan Gwang Yeogsi
  - Yeungnam University Medical Center /ID# 269992, Daegu
  - Seoul Songdo Hospital /ID# 270009, Junggu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-081